CLINICAL TRIAL: NCT05138679
Title: Prospective Multicenter Observational Study Evaluating Acute Lower Limb Ischemia
Brief Title: Evaluation of Acute Lower Limb Ischemia
Acronym: PROMOTE-ALI
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1220/2021
Record Dates: First submitted 2021-11-15; First posted 2021-12-01 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2021-08

CONDITIONS: Acute Limb Ischemia
Keywords: acute lower limb ischemia; revascularization; compartment syndrome; limb salvage; COVID-19
MeSH Terms: conditions — Compartment Syndromes; COVID-19 | interventions — Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute lower limb ischemia: Patients with acute lower limb ischemia (older than 18 years)
  Interventions: Procedure: Revascularization; Procedure: Primary major amputation; Other: Best medical treatment

INTERVENTIONS:
Procedure: Revascularization — Endovascular or surgical restoration of arterial blood flow.
  Other Names: Surgical embolectomy; Peripheral bypass; Catheter directed thrombolysis; Catheter guided aspiration; Catheter guided atherectomy; Percutaneous transluminal angioplasty
Procedure: Primary major amputation — Primary below- or above knee major amputation without prior revascularization.
Other: Best medical treatment — Conservative treatment of acute lower limb ischemia - without prior revascularization.

SUMMARY:
The primary objective of this study is to evaluate the effect of different treatment modalities on clinical outcome of patients suffering from acute lower limb ischemia (ALI). Depending on clinical presentation, anatomical as well as technical considerations, different treatment options are available for revascularisation of affected limbs. Using an observational, international, multicentric study design (min. patient number of 500), the defined primary endpoint of the study, amputation-free survival 90 days after the diagnosis of ALI, will be evaluated.

DETAILED DESCRIPTION:
Recently published clinical guidelines highlighted that the available evidence on the management of acute lower limb ischemia (ALI) is mostly outdated and includes only small patient cohorts. Depending on the patient's characteristics, the duration of ischemic symptoms as well as the cause of ALI and the anatomical lesion, different treatment options are available and need to be compared regarding clinical outcome.

With the knowledge about the heterogeneity of patients suffering from ALI, a multicentre observational study design has the potential to give results on influence of several factors (patient related factors, treatment related factors) on clinical outcome of patients with lower extremity ALI. In contrast, a randomized controlled trial would not be feasible as heterogeneity of patients would lead to limitations in the recruitment of patients.

The primary objective of this study is to evaluate the effect of different treatment modalities on clinical outcome of patients suffering from acutle lower limb ischemia. Depending on clinical presentation, anatomical as well as technical considerations, different treatment options are available for revascularisation of affected limbs. Using an observational, international, multicentric study design (min. patient number of 500), the defined primary endpoint of the study, amputation-free survival 90 days after the diagnosis of ALI, will be evaluated.

The secondary objectives of this study are the identification of factors having an effect on the primary endpoint . These factors are:

* Demographic data (age, gender, Body Mass Index,
* Cardiovascular risk factors (diabetes, arterial hypertension, dyslipidemia, smoking history)
* COVID-19 anamnesis (infectious status; vaccination status)
* Pre-existing diseases (Arterial fibrillation, chronic kidney disease, hemodialysis, coronary artery disease, COVID infection in medical history, pulmonary disease)
* Risk factors for ALI (peripheral arterial disease, aortic aneurysm or dissection, arterial embolization in medical history, malignant disease, peripheral arterial aneurysm, previous stroke, thrombophilia, revascularization procedure on ipsilateral limb)
* Pre-existing medication (antiplatelet, oral anticoagulation, statins)
* Clinical presentation (Rutherford ischemia classification, Cause of ALI, anatomical level of arterial occlusion, diagnostic imaging modality)
* Details on performed intervention (time of ischemia, periprocedural heparin administration, type of procedure, technical details on performed procedure, compartment syndrome with need for fasciotomy)
* Outcome parameters (Survival, Rutherford ischemia classification, residual sensory or motor deficit, impaired walking distance, need for reintervention, major bleeding periprocedural, access site complications, organ failure) 30 and 90 days after diagnosis of ALI.

ELIGIBILITY:
Inclusion Criteria:

* Acute lower limb ischemia (Rutherford Categories I-III)

Exclusion Criteria:

* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with the diagnosis of acute lower limb ischemia treated at a participating study center.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Amputation free survival - rate | 90 days
  Rate of amputation free survival after diagnosis of acute lower limb ischemia

SECONDARY OUTCOMES:
Re-intervention rate of the index leg | 90 days
  Rate of re-intervention for revascularization or complications of the index-leg
Complication rate | 90 days
  Rate of complications after the diagnosis of acute limb ischemia (access site infection, acute kidney injury, periprocedural major bleeding, compartment syndrome, multi organ failure)
Limb salvage rate | 90 days
  Rate of patients not requiring major amputation.
Survival rate | 90 days
  Rate of patients surviving the diagnosis of acute limb ischemia until the end of follow-up
Clinical outcome of the index leg (Rutherford category) | 90 days
  Clinical symptoms at the end of follow up (Rutherford category)

CONTACTS AND LOCATIONS:
Overall Officials: Florian K Enzmann, MD, PhD, Principal Investigator — Department of Vascular Surgery, Medical University of Innsbruck; Alexandra Gratl, MD, Principal Investigator — Department of Vascular Surgery, Medical University of Innsbruck
Locations (37):
- Austria (4):
  - Medical University of Innsbruck, Department of Vascular Surgery, Innsbruck
  - Department of General Surgery, Division of Vascular Surgery, Medical University of Vienna, Vienna
  - Department of Vascular and Endovascular Surgery, Hospital Ottakring, Vienna
  - Department of Cardio-Vascular Surgery, Clinic Floridsdorf and Karl Landsteiner Institute for Cardio-Vascular Research, Vienna
- University Hospital Merkur, Zagreb, Croatia
- France (15):
  - Department of Vascular Surgery, Hospital of Antibes Juan-les-Pins, Antibes
  - Department of Vascular Surgery, Bordeaux University Hospital, Bordeaux
  - Department of Vascular Surgery, Ambroise Paré University Hospital, Assistance Publique-Hôpitaux de Paris, Boulogne-Billancourt
  - Department of Vascular and Endovascular Surgery, Brest University Hospital, Brest
  - Department of Vascular Surgery, Henri Mondor University Hospital, Créteil
  - Department of Vascular Surgery, University Hospital of Dijon, Dijon
  - Vascular Surgery Department, Hospices Civils de Lyon, Lyon
  - Department of Vascular Surgery, University Hospital of Nancy, Nancy
  - CHU Nantes, l'institut du thorax, service de chirurgie cardio-vasculaire, Nantes
  - University Hospital of Nice, Université Côte d'Azur, Nice
  - Department of Vascular and Thoracic Surgery, Bichat Hospital, Paris, Université de Paris, Paris
  - Department of Vascular Surgery, Ambroise Paré University Hospital, Boulogne-Billancourt and Simone Veil Health Sciences Medical School, Versailles-Saint-Quentin-en-Yvelines University and Paris-Saclay University, Paris
  - Vascular Surgery Department, Georges Pompidou European Hospital, APHP, Paris University, Paris
  - Department of Vascular Surgery, CHU de Reims, Reims
  - Department of Vascular Surgery and Kidney Transplantation, University Hospitals of Strasbourg, Strasbourg
- Germany (5):
  - European Vascular Center Aachen-Maastricht, University Hospital Aachen, RWTH Aachen University, Aachen
  - University Hospital Cologne, Cologne
  - Division of Vascular and Endovascular Surgery Department for Visceral-, Thoracic and Vascular Surgery Medical Faculty Carl Gustav Carus and University Hospital Carl Gustav Carus Dresden Technische Universität Dresden, Dresden
  - Department of Vascular- and Endovascular Surgery, Medical Faculty and University Hospital Düsseldorf, Heinrich-Heine-University Düsseldorf, Düsseldorf
  - Department of Vascular and Endovascular Surgery, University Hospital Münster, Münster
- Department of Vascular and Endovascular Surgery, Heart and Vascular Center, Semmelweis University, Budapest, Hungary
- University Hopspital Chișinău, Chisinau, Moldova
- Netherlands (2):
  - Amsterdam University Medical Center, Department of Surgery, Amsterdam
  - University Medical Center Utrecht, Department of Vascular Surgery, Utrecht
- Serbia (3):
  - Clinic for Vascular and Endovascular Surgery, Clinical Center of Serbia, Belgrade
  - Institute for Cardiovascular Disease, Belgrade, Belgrade
  - Clinic for Vascular Surgery, Clinical Center Niš, Niš
- Switzerland (2):
  - Department of Cardiovascular Surgery, Inselspital, University of Bern, Bern
  - Department of Vascular Surgery, Kantonsspital Winterthur, Winterthur
- United Kingdom (3):
  - Bristol Centre for Surgical Research, Bristol NIHR Biomedical Research Centre, University of Bristol, Bristol
  - Department of Vascular Surgery, University Hospital Wales, Cardiff
  - NHS Lothian, Edinburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behrendt CA, Bjorck M, Schwaneberg T, Debus ES, Cronenwett J, Sigvant B; Acute Limb Ischaemia Collaborators. Editor's Choice - Recommendations for Registry Data Collection for Revascularisations of Acute Limb Ischaemia: A Delphi Consensus from the International Consortium of Vascular Registries. Eur J Vasc Endovasc Surg. 2019 Jun;57(6):816-821. doi: 10.1016/j.ejvs.2019.02.023. Epub 2019 May 22. PMID 31128987
- [Background] Bjorck M, Earnshaw JJ, Acosta S, Bastos Goncalves F, Cochennec F, Debus ES, Hinchliffe R, Jongkind V, Koelemay MJW, Menyhei G, Svetlikov AV, Tshomba Y, Van Den Berg JC, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Kakkos SK, Koncar I, Lindholt JS, Tulamo R, Vega de Ceniga M, Vermassen F, Document Reviewers, Boyle JR, Mani K, Azuma N, Choke ETC, Cohnert TU, Fitridge RA, Forbes TL, Hamady MS, Munoz A, Muller-Hulsbeck S, Rai K. Editor's Choice - European Society for Vascular Surgery (ESVS) 2020 Clinical Practice Guidelines on the Management of Acute Limb Ischaemia. Eur J Vasc Endovasc Surg. 2020 Feb;59(2):173-218. doi: 10.1016/j.ejvs.2019.09.006. Epub 2019 Dec 31. No abstract available. PMID 31899099
- [Derived] Gratl A; European Vascular Research Collaborative (EVRC). Study Protocol of a Prospective Multicenter Observational Study Evaluating Acute Lower Limb Ischemia. J Surg Res. 2023 Feb;282:280-284. doi: 10.1016/j.jss.2022.09.023. Epub 2022 Nov 5. PMID 36347128